CLINICAL TRIAL: NCT00626444
Title: Phase II Trial of High Dose Intravenous Vitamin C in Patients With Refractory Non-Hodgkin Lymphoma
Brief Title: Pilot Trial of Intravenous Vitamin C in Refractory Non-Hodgkin Lymphoma (NHL)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Responsible Party: Sponsor
Organization: Thomas Jefferson University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07U.21; JT 1201 (Other: JeffTrial Number)
Record Dates: First submitted 2008-02-21; First posted 2008-02-29 (Estimated); Results first posted 2014-12-10 (Estimated); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Non-Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Intravenous vitamin C
  Interventions: Drug: Intravenous vitamin C

INTERVENTIONS:
Drug: Intravenous vitamin C — Up to 100 gms of intravenous vitamin C, three times per week for 10 weeks.

SUMMARY:
Eligible candidates will be adults with aggressive or very aggressive NHL (WHO classification diagnosis confirmed by histological tumor examination). Patients must have failed one or more prior NHL chemotherapy or antibody therapy with curative intent, and the disease must not have progressed within 60 days of last therapy. In addition, patients must not be candidates for potentially curative therapy, such as HSCT, or they must have refused these alternative therapies. Full inclusion/exclusion criteria are available. History and physical examination, and laboratory and imaging analyses will be done within 14 days prior to registration. Intravenous ascorbic acid will be given in a dose based on the plasma vitamin C level to reach a level in the range of 300 to 350 mg/dL. Vitamin C infusions will be given three times a week on a schedule that allows at least 24 hours between each infusion, for a total of ten weeks (30 infusions). If disease progression occurs before or at the ten week assessment, then we discontinue protocol, based on futility. Toxicity and adverse events also will result in immediate discontinuation (details available in full protocol). If there is lack of disease progression or disease improvement, proceed and reassess again at 10 week intervals, for a total of three 10 week intervals. Initial criteria are based upon the criteria from the International Workshop to Standardize Criteria for Non-Hodgkin's Lymphoma (Cheson et al., Report of an international workshop to standardize response criteria for non-Hodgkin's lymphoma, Journal of Clinical Oncology, 1999, Vol. 17, No4, 1244-1253); response for this study will utilize PET in accordance with revised criteria (Cheson et al. Revised response criteria for malignant lymphoma. J of Clin Oncol 2007; 25(5): 579-586). We select 20 patients as an appropriate study size to evaluate a true response rate to therapy, compared to just the observed response.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18 years old
* Aggressive or very aggressive NHL
* Failed one or more therapies
* Patients must not have progressed within 60 days of last therapy
* Not received allogeneic stem cell transplant
* No reasonable standard therapeutic options available
* Glucose 6 phosphate dehydrogenase status normal
* ECOG performance status 0-2
* Normal creatinine and transaminase
* Women of child-bearing potential confirm negative pregnancy test

Exclusion Criteria:

* Significant co-morbid disorders
* Significant psychiatric symptoms
* Smoking
* Excessive alcohol or drug use
* Enrollment in other experimental therapy
* Active infection
* Patients experiencing ongoing response to recent treatments
* Patients who have received chemotherapy within 30 days or biological therapy within 6 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2008-02; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Monti, MD, Principal Investigator — Faculty Member
Locations (1):
- Jefferson-Myrna Brind Center of Integrative Medicine, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Vitamin C: Intravenous vitamin C
  Intravenous vitamin C: Up to 100 gms of intravenous vitamin C, three times per week for 10 weeks.
Period: Overall Study
Arm/Group | Vitamin C
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Vitamin C
Number analyzed (Participants) | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.3 (2.9)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Time Frame: 10 weeks
Arm/Group | Vitamin C
Number analyzed (Participants) | 0

2. Secondary Outcome: Duration of Response
Time Frame: 10 weeks
Arm/Group | Vitamin C
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Vitamin C
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 2/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vitamin C (N=2)
Abdominal pain (General disorders) | 1 (1)
Back pain (General disorders) | 1 (1)
Induration at IV site (General disorders) | 1 (1)
Lightheadedness (General disorders) | 1 (1)
Nausea (General disorders) | 1 (1)
Pain at IV site (General disorders) | 1 (3)
Viral illness (General disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Study was terminated due to poor accrual. No reportable data has been collected for any of the specified outcome measures.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes